CLINICAL TRIAL: NCT04410809
Title: A SINGLE-CENTER, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP STUDY INVESTIGATING THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF SINGLE- AND MULTIPLE-ASCENDING SUBCUTANEOUS DOSES OF TA-46 IN HEALTHY VOLUNTEERS
Brief Title: Study Of Safety, Tolerability And Pharmacokinetics Of Subcutaneous Doses Of TA-46
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TA46-001; 2017-003596-55 (EudraCT Number); C4181002 (Other: Alias Study Number)
Record Dates: First submitted 2020-05-28; First posted 2020-06-01 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): The same composition as the active medication but without the active substance TA-46
  Interventions: Other: Placebo
- TA-46 (Experimental): Decoy protein of the fibroblast growth factor receptor 3
  Interventions: Biological: TA-46

INTERVENTIONS:
Biological: TA-46 — Decoy protein of the fibroblast growth factor receptor 3, 50 mg/mL (Parts A, B and C) and 120 mg/mL (Part C and Part D), sc solution for injection/infusion
  Arms: TA-46
Other: Placebo — The same composition as the active medication but without the active substance TA-46
  Arms: Placebo

SUMMARY:
TA-46 single- and multiple-ascending dose study in healthy volunteers to investigate safety and PK. The protocol is conducted in four parts; Part A - Single Ascending doses of TA46 Part B - Multiple Ascending doses of TA-46 Part C - Comparing 2 formulations 50mg/ml vs 120mg/ml TA-46 Part D - Single Ascending dose of TA46 120mg/ml formulation

The subjects will be in the clinic for 1 period. The subjects will be admitted to the clinical research center in the afternoon of Day -1. They will be discharged on Day 4 (72 hours post-dose) after completion of the assessments. After discharge, the subjects will return to the clinical research center for ambulatory visits on Days 5, 8, 10, 12, 14 and 22

DETAILED DESCRIPTION:
This is a single-center, 34-part clinical study in healthy subjects.

Part A This is a single-center, double-blind, randomized, placebo-controlled, single ascending dose study in healthy subjects. The dose escalation is adaptive in nature. An estimated number of 5 dose levels will be administered in Part A of the study, with at each dose level 6 subjects randomized to receive TA-46 and 2 to receive placebo. Depending on evaluation of the data the number of subjects may be adjusted and/or additional group(s) may be added.

In this first-in-human study, the subjects participating at all dose levels of Part A (Groups A1-A5), will be dosed according to a sentinel dosing design to ensure optimal safety. This means that initially 2 subjects will be dosed: 1 subject with TA-46 and 1 subject with placebo. If the safety and tolerability results of the first 24 hours following dosing for the initial subjects are acceptable to the Principal Investigator (PI), the other 6 subjects (5 active and 1 placebo) of that dose level may be dosed.

For Groups A1 and A2, TA-46 and placebo will be administered as a sc injection (bolus) and for Groups A3-A5, TA-46 and placebo will be administered as a sc infusion. When TA-46 and placebo will be administered as sc infusion, the duration of the sc infusion will be dependent on the volume to be administered, but will not exceed a period of 1 hour. The dose levels of TA-46 can be increased or decreased based on the results of the previous group(s).

Part B This is a single-center, double-blind, randomized, placebo-controlled, multiple ascending dose study in healthy subjects. The dose escalation is adaptive in nature. TA-46 will be administered twice weekly for4 weeks. An estimated number of 3 dose levels will be administered in Part B of the study, with at each dose level 6 subjects randomized to receive TA-46 and 2 to receive placebo. Depending on evaluation of the data the number of subjects may be adjusted and/or additional group(s) may be added. Based on the results of Groups B1 and B2 of Part B, which followed a twice weekly dosing scheme for 4 weeks, the dosing scheme of Group B3 will be adapted to once weekly administration for 4 weeks and 31 additional groups (Groups B4 to B6) with the same dosing frequency will be added to Part B of the study. Depending on evaluation of the data, additional group(s) may be added or planned group(s) may be skipped.

For Group B1, TA-46 and placebo will be administered as a sc injection (bolus) and for Groups B2 to B64, TA-46 and placebo will be administered as a sc infusion. When TA-46 and placebo will be administered as a sc infusion, the duration of the sc infusion will be dependent on the volume to be administered, but will not exceed a period of 1 hour. The dose levels of TA-46 can be increased or decreased based on the results of the previous group(s).

Administration of a dose level in Part B can be started after completion and review of the corresponding or higher dose level in Part A of the study.

Part C This is a single-center, single-dose, open-label, cross-over study in healthy subjects comparing 2 formulations of TA-46 (50 mg/mL and 120 mg/mL). A total of 6 subjects will receive Treatment A (TA-46 formulation 1) and Treatment B (TA-46 formulation 2) randomly assigned over 2 periods with 2 treatment sequences (Treatment A/B and Treatment B/A) with 3 subjects per treatment in each sequence.

The following treatments are planned to be administered according to the randomization code:

Group C1 Treatment A: sc administration of 3 mg/kg TA-46 formulation 1 Treatment B: sc administration of 3 mg/kg TA-46 formulation 2TA-46 formulation 1 will be administered as a a sc infusion. The duration of the sc infusion will be dependent on the volume to be administered, but will not exceed a period of 1 hour. TA-46 formulation 2 will be administered as 1-2 sc injection(s) (bolus).

The subjects will be in the clinic for 2 periods. Each period the subjects will be admitted to the clinical research center in the afternoon of Day -1 and they will be discharged on Day 4 (72 hours post-dose) after completion of the assessments. After discharge, the subjects will return to the clinical research center for ambulatory visits on Days 6, 9, 12, 16, and 22 of each period.

Part D This is a single-center, open-label, single-dose study in healthy subjects with the TA-46 formulation of 120 mg/mL.

TA-46 and placebo will be administered as a sc infusion. The duration of the sc infusion will be dependent on the volume to be administered, but will not exceed a period of 1 hour. Depending on evaluation of the data, additional group(s) may be added or planned group(s) may be skipped.

ELIGIBILITY:
Inclusion Criteria:-

* Age : 21-55 years, inclusive, at screening
* Weight : maximum weight of 100 kg
* Normal height without any growth complications during childhood
* Healthy as determined by screening assessments

Exclusion Criteria:

* Concomitant disease or condition that could interfere with, or for which the treatment might interfere with, the conduct of the study, or that would, in the opinion of the PI, pose an unacceptable risk to the subject in this study
* Clinically significant abnormalities in laboratory test results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis)
* Participation in an investigational drug or device study within 3 months prior to (the first) drug administration in the current study

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Bsseline to Day 43 after last dose of study medication
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Y days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug X was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of Participants With Clinical Laboratory Abnormalities | Baseline up to Day 43 after last dose of study medication
  Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); liver function (aspartate aminotransferase, alanine aminotransferase, total bilirubin, lactate dehydrogenase, alkaline phosphatase, albumin, total protein); renal function (blood urea nitrogen, creatinine, uric acid); electrolytes (sodium, potassium, chloride, calcium, phosphate, bicarbonate); clinical chemistry (glucose, creatine kinase); immunology (CRP); urinalysis (dipstick [urine specific gravity, decimal logarithm of reciprocal of hydrogen ion activity {pH} of urine, glucose, protein, blood, ketones, bilirubin], microscopy [urine RBC, WBC, urate crystals, calcium, oxalate, miscellaneous [urine mucus and leucocytes]).
Incidence of Anti-Drug Antibody (ADA) | Baselin up to Day 43 after last dose of study medication
  The percentage of participants with positive ADA and neutralizing antibodies will be summarized for each treatment arm.
Number of Participants With Change From Baseline in Physical Examinations and Vital Signs | Baseline up to Day 43 after last dose study medication
  Number of participants with potentially clinically important (PCI) physical examinations and vital signs is reported during therapy and at post therapy. Criteria for PCI change in vital signs: heart rate value of <40 beats per minute and value >150 beats per minute, systolic blood pressure (SBP) of <80 or >210 millimeter of mercury (mmHg), diastolic blood pressure (DBP) of <40 or >130 mmHg, temperature <32 or >40 degree centigrade, respiratory rate of <10 or >50 breaths/minute and criteria for PCI change in physical examination: >=10% increase or decrease of body weight in kilogram (kg).
Number of Participants With Abnormal Electrocardiogram (ECG) | Baseline up to Day 22 after last dose of study medication
  Criteria for ECG abnormalities: maximum PR interval >=300 milliseconds (msec) and maximum increase PR interval increase from baseline (IFB): percent change (Pctchg) >=25 percent (%) for baseline value of >200 msec and Pctchg>=50% for baseline value of <=200 msec for PR interval, maximum QRS interval >=140 msec and a maximum IFB: Pctchg>=50%, maximum QTCF interval (Fridericia's Correction) of 450 msec to <480 msec, 480 msec to <500 msec or >=500 msec and a maximum change of <=30change<60 or >=60 msec from baseline.

SECONDARY OUTCOMES:
Area under the Concentration-Time Curve (AUC) | BaselineDay 1, Day , Day 15, Day 22 & Day 25, Day 29 post dose
  AUC is a measure of the serum concentration of the drug over time. It is used to characterize drug absorption.
Cmax | Baseline, Day 1, Day , Day 15, Day 22 & Day 25, Day 29 post dose
  To compare the safety, tolerability and PK of single sc doses of 2 formulations of TA-46 (50 mg/mL and 120 mg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PRA, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=TA46-001